CLINICAL TRIAL: NCT05451797
Title: A Feasibility Study Into the Implant of the WiSE CRT System With an Intracardiac Pacemaker to Achieve Totally Leadless CRT
Brief Title: Implant of the WiSE CRT System With an Intracardiac Pacemaker
Acronym: TLC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: EBR Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DEV DVD0024
Record Dates: First submitted 2022-06-12; First posted 2022-07-11 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Implant of WiSE-CRT with intracardiac pacemaker — Implant of two cardiac devices

SUMMARY:
This study is a single arm, prospective, feasibility, multi-centre, observational study. Participants will be suitable for a Cardiac Resynchronisation Therapy (CRT) implant using Wireless Stimulation Endocardially for Cardiac Resynchronization Therapy, known as the WiSE-CRT device system as well as requiring a pacemaker implant which will also be leadless. Some of these participants may also require an AV Node ablation.

The purpose of this study is to assess the safety and efficacy of these two cardiac devices implanted in the order of operator preference (all implants undertaken on the same day or in a number of up to 4 separate sequenced implants/procedures).

DETAILED DESCRIPTION:
Heart Failure is a serious condition in which the heart is unable to pump enough blood to meet the body's demands. Some heart failure occurs when the heart chambers pump in a desynchronised manner, reducing the amount of blood pumped with each heartbeat.

The National Institute for Health and Care Excellence (NICE) recommends Cardiac Resynchronisation Therapy (CRT) for a subset of these patients. Patients undergoing CRT receive a special implantable pacemaker with an additional lead via the coronary sinus (CS) to synchronise the pumping of the heart chambers (ventricles). CRT works by pacing both the left & right ventricles to ensure they pump at the same time. This in turn, reduces heart failure symptoms.

CRT is an effective treatment for many patients, but limitations prevent some patients from benefiting:

* 5-10% of patients are considered untreated due to acute/chronic issues with the CS lead
* 30% of patients do not respond/improve

The WiSE-CRT System is an implantable pacing system capable of delivering pacing energy to the heart without using a pacing lead. It was designed to address the persistent limitations of current CRT systems. The WiSE-CRT System operates alongside a co-implanted pacemaker or CRT system and replaces the pacing function of the CS lead.

Intracardiac pacemakers are miniaturized, self-contained, pacing systems implanted directly inside the right ventricle of the heart, eliminating the need for a device pocket and pacing lead inserted into a vein.

By co-implanting both the European conformity certificated (CE marked) WiSE-CRT system and a leadless intracardiac pacemaker, this pilot study will assess the safety and efficacy of implanting a totally leadless system, thereby avoiding both acute and chronic complications associated with the implant of transvenous pacing leads.

This study is a single arm, prospective, multi-centre, observational study. Participants will have initial pre-implant screening baseline measurements prior to implantation of the first system, then will be followed up immediately post implant, then at 1 month & 6 months post implant.

ELIGIBILITY:
Inclusion Criteria:

Male or Female, aged 18 years or above. Participant is willing and able to give informed consent for participation in the study.

Additionally, participants will be enrolled and classified from one of two distinct groups:

GROUP A: De novo totally leadless CRT

* implant in whom the physician believes a totally leadless approach would be beneficial (e.g. wish to avoid lifelong transvenous lead implant, anatomical constraints, history of device infection). Examples of this could include:
* symptomatic atrial fibrillation (AF) and an uncontrolled heart rate who are candidates for AV node ablation (irrespective of QRS duration and ejection fraction), in whom the physician believes a leadless pacing approach would be beneficial.
* high degree atrioventricular block who has an indication for permanent pacing, with an ejection fraction ≤50%, are expected to require ventricular pacing more than 40% of the time and in whom the physician believes a leadless approach would be beneficial.
* Other indications for leadless pacing including venous obstruction, pocket issues, infection risk (eg: chronic dialysis), etc.

GROUP B: Upgrade chronic intracardiac pacemaker to CRT

o Patient with existing intracardiac pacemaker with greater than 20% right ventricular (RV) pacing, who have developed symptomatic heart failure.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the study
* Inability to comply with the study follow-up or other study requirements
* History of chronic alcohol/drug abuse and currently using alcohol/drugs
* Non-ambulatory (or unstable) NYHA class 4
* Life expectancy less than 12 months
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Enrolled in another clinical study that could confound the results of this study (note: patients enrolled in complementary study are eligible for enrolment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients appropriate for these devices
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety from major complications post device implants & procedures | 6 months
  Freedom from major complications following device implants and procedures, whether single stage or multiple staged procedures. Major complications are defined as any complication related to the device or procedure that results in death, hospitalization, prolongation of hospitalisation for 48 or more hours, permanent loss of device function due to a mechanical or electrical malfunction or system change (removal, repositioning, or replacement).
Efficacy of Cardiac Resynchronisation Therapy (CRT) measured by confirmation of Bi Ventricular Pacing on 12 lead ECG. | 6 months
  Evidence of biventricular pacing on 12 lead ECG recorded at 6 months will confirm CRT delivered by implanted devices for each participant.

SECONDARY OUTCOMES:
Clinical Response of Each Participant measuring Left Ventricular Ejection Fraction. | 6 months
  This will be measured by using a recognised clinical tool that reflects the participant's heart failure status by measuring the left ventricular contractility of the heart. Changes at 6 months (relative to baseline measurement) in Left Ventricular Ejection Fraction as a % from Transthoracic Echocardiogram (TTE) will be measured.
Clinical Response of Each Participant measuring Left Ventricular End Systolic Volume. | 6 months
  Changes at 6 months (relative to baseline measurement) in Left Ventricular End Systolic Volume in ml on Transthoracic Echocardiogram. This is a recognised clinical tool that reflects the participant's heart failure status by measuring the left ventricular contractility of the heart.
Clinical response of Each Participant measuring New York Heart Association classification. | 6 months
  Changes at 6 months (relative to baseline measurement) in New York Heart Association classification (class I, II, III or IV). This is a recognised clinical tool that reflects the participant's heart failure status. Class I is least severe and reflects no physical symptoms whilst under going normal physical activity through to class IV, most severe, and unable to carry out any physical activity without discomfort and may have symptoms at rest.
Clinical response of Each Participant measuring 6 Minute Walk Test | 6 months
  Changes at 6 months (relative to baseline measurement) in 6 minute walk test measured in metres. This is a recognised clinical tool that reflects the Participant's heart failure status by measuring how far the participant can walk during a 6 minute period on flat terrain.

OTHER OUTCOMES:
Analysis of single stage and multiple stage device implant procedure times | 6 months
  Comparing mean procedural times of single stage device implants, or up to 4 stage implant procedure times, as per operator preference.

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Roberts, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No